CLINICAL TRIAL: NCT01002300
Title: Investigation of the Effects of Intranasal Oxytocin on Cognition and Emotion Processing in Frontotemporal Dementia
Brief Title: Oxytocin and Social Cognition in Frontotemporal Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: The Alzheimer Society London and Middlesex (Other)
Responsible Party: Principal Investigator, Elizabeth Finger, Cognitive Neurologist, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R-08-395; 15398
Record Dates: First submitted 2009-10-23; First posted 2009-10-27 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Frontotemporal Dementia; Pick's Disease
Keywords: Social Cognition; Oxytocin
MeSH Terms: conditions — Frontotemporal Dementia; Pick Disease of the Brain | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: intranasal oxytocin — Participants will receive 24 IU of oxytocin or placebo (Salinex saline nasal spray) intranasally 30 minutes prior to completing the experimental tasks. Two weeks later participants will return for a second visit and receive the alternate drug (either intranasal oxytocin or Salinex) prior to completing the experimental tasks.
  Other Names: Syntocinon

SUMMARY:
Investigations into the components of cognition damaged in frontotemporal dementia (FTD) demonstrate that patients with FTD show deficits in facial and verbal expression recognition, lack insight into what others think or might do (theory of mind skills), and in decision making tasks requiring processing of positive versus negative feedback. These cognitive functions are thought to be critical for appropriate social behavioural regulation (Blair, 2003). Recent studies in animal models and humans suggest that the neuropeptide oxytocin is an important mediator of social behavior and that oxytocin may facilitate emotion recognition, theory of mind processing, and prosocial behaviors (Donaldson and Young, 2008). Together, these findings suggest that upregulation of oxytocin dependent mechanisms of social and emotional cognition may be a valuable treatment approach in patients with FTD. The aim of this study is to determine how administration of intranasal oxytocin to patients with frontotemporal dementia affects behavior and processing of specific types of social and emotional information.The investigators' hypothesis is that oxytocin administration will improve emotional and social cognitive deficits in patients with FTD, resulting in improved decision making and behaviour.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of probable Frontotemporal Dementia or Pick's disease
* Caregiver available to participate in all study visits

Exclusion Criteria:

* Severe language or memory deficits that preclude completion of the cognitive tasks
* Females who are pregnant or breastfeeding (a pregnancy test will be done on females who have not completed menopause)
* Uncontrolled hypertension
* Bradycardia (rate <50 bpm) or tachycardia (rate > 100 bpm)
* Current use of prostaglandins
* Use of any investigational or experimental drug or device within the last 60 days prior to screening or within 5 half-lives of the experimental drug , whichever is longer

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Performance on Emotion Recognition Tasks | Day of treatment

SECONDARY OUTCOMES:
Behavioural Ratings of Emotional Sensitivity and Repetitive Behaviours | One week following treatment
Side effects | 1 week after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth C Finger, MD, Principal Investigator — University of Western Ontario/ St. Joseph's Hospital, Lawson Research Institute
Locations (1):
- Cognitive Neurology and Alzheimer's Research Centre, St. Joseph's Hospital, London, Ontario, Canada

REFERENCES:
- [Background] Guastella AJ, Mitchell PB, Dadds MR. Oxytocin increases gaze to the eye region of human faces. Biol Psychiatry. 2008 Jan 1;63(1):3-5. doi: 10.1016/j.biopsych.2007.06.026. Epub 2007 Sep 21. PMID 17888410
- [Background] Donaldson ZR, Young LJ. Oxytocin, vasopressin, and the neurogenetics of sociality. Science. 2008 Nov 7;322(5903):900-4. doi: 10.1126/science.1158668. PMID 18988842
- [Background] Hollander E, Bartz J, Chaplin W, Phillips A, Sumner J, Soorya L, Anagnostou E, Wasserman S. Oxytocin increases retention of social cognition in autism. Biol Psychiatry. 2007 Feb 15;61(4):498-503. doi: 10.1016/j.biopsych.2006.05.030. Epub 2006 Aug 14. PMID 16904652